CLINICAL TRIAL: NCT03361007
Title: Evaluation of Clinical Outcomes of Transcatheter Aortic Valve Implantation Through Common Carotid Artery Access in Polish Population - Observational Multicenter Registry
Brief Title: Polish Registry of Common Carotid Artery Access for TAVI
Acronym: POL-CAROTID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: WUM-CCA
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Aortic Valve Stenosis; Ventricular Outflow Obstruction, Left
Keywords: TAVI; common carotid artery
MeSH Terms: conditions — Aortic Valve Stenosis; Ventricular Outflow Obstruction, Left | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Common carotid artery access for TAVI: Patients in whom femoral artery could not be used to deliver the bioprosthesis for any reason.
  Interventions: Device: Transcatheter Aortic Valve Implantation (TAVI)

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation (TAVI) — Patients who were disqualified from surgical cortical valve replacement by decision of the Heart Team.
  Other Names: Transcatheter Aortic Valve Replacement (TAVR)

SUMMARY:
Transcatheter aortic valve implantation (TAVI) is valuable treatment option for patients, who are at the high risk of surgical aortic valve replacement (AVR). Majority of procedures are performed through femoral arteries, however in some this access cannot be applied. Common carotid artery is one of the alternative routes of delivering the device in those patients. Established registry aims at collecting the data prospectively to assess outcomes of TAVI through common carotid artery.

DETAILED DESCRIPTION:
The study is a prospective multicenter evaluation of transcatheter aortic valve implantations through common carotid artery in Polish health centers.

Duration of this study is expected to be 6 years to ensure that all of the enrolled patients will complete at least 2 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Qualification for TAVI through common carotid artery by decision of the local Heart Team
* Patient provided written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients meeting inclusion criteria will prospectively included in the study. Patients meeting inclusion criteria before the set-up of registry will be included retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
VARC (Valve Academic Research Consortium-2) defined "Clinical Efficacy" composite endpoint | From 30 days post procedure to completion of at least 2 years of follow up
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Requiring hospitalizations for valve-related symptoms or worsening congestive heart failure
  * NYHA (New York Heart Association) class III or IV functional classification of heart failure
  * Valve-related dysfunction (mean aortic valve gradient ≥20 mmHg, Effective Orifice Area (EOA) ≤0.9-1.1 cm2(c) and/or Doppler Velocity Integral (DVI) <0. 35 m/s, AND/OR moderate or severe prosthetic valve regurgitation

SECONDARY OUTCOMES:
VARC defined 'Device success' composite endpoint | 30 days
  * Absence of procedural mortality AND
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location AND
  * Intended performance of the prosthetic heart valve (no prosthesis - patient mismatch and mean aortic valve gradient ,20 mmHg or peak velocity ,3 m/s, AND no moderate or severe prosthetic valve regurgitation)
VARC defined "Early Safety" composite endpoint | 30 days
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening bleeding
  * Acute kidney injury-Stage 2 or 3 (including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complication
  * Valve-related dysfunction requiring repeat procedure (Balloon Aortic Valvuloplasty (BAV), Trans Catheter Aortic Valve Implant (TAVI), or Surgical Aortic Valve Replacement (SAVR))
VARC defined "Time-related valve safety" composite endpoint | From device implant to completion of at least 2 years of follow up
  * Structural valve deterioration
  * Valve-related dysfunction (mean aortic valve gradient ≥20 mmHg, EOA ≤0.9-1.1 cm2cand/or DVI <0.35 m/s, AND/OR moderate or severe prosthetic valve regurgitation)
  * Requiring repeat procedure (TAVI or SAVR)
  * Prosthetic valve endocarditis
  * Prosthetic valve thrombosis
  * Thrombo-embolic events (e.g. stroke)
  * VARC bleeding, unless clearly unrelated to valve therapy (e.g. trauma)

CONTACTS AND LOCATIONS:
Overall Officials: Zenon Huczek, MD, PhD, Principal Investigator — Medical University of Warsaw; Radosław Wilimski, MD, Principal Investigator — Medical University of Warsaw
Locations (6):
- Poland (6):
  - Medical University of Gdansk, Gdansk
  - Medical University of Silesia, Katowice
  - Medical University of Lodz, Lodz
  - University of Opole, Opole
  - Poznan University of Medical Sciences, Poznan
  - Medical University of Warsaw, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huczek Z, Wilimski R, Kochman J, Szczudlik P, Scislo P, Rymuza B, Kaplon-Cieslicka A, Kolasa A, Marchel M, Filipiak KJ, Cichon R, Opolski G. Common carotid artery access for transcatheter aortic valve implantation. Kardiol Pol. 2015;73(7):478-84. doi: 10.5603/KP.2015.0122. PMID 26189468
- [Background] Azmoun A, Amabile N, Ramadan R, Ghostine S, Caussin C, Fradi S, Raoux F, Brenot P, Nottin R, Deleuze P. Transcatheter aortic valve implantation through carotid artery access under local anaesthesia. Eur J Cardiothorac Surg. 2014 Oct;46(4):693-8; discussion 698. doi: 10.1093/ejcts/ezt619. Epub 2014 Jan 14. PMID 24431170
- [Background] Schirmer J, Conradi L, Seiffert M, Koschyk D, Blankenberg S, Reichenspurner H, Diemert P, Treede H. Transcatheter aortic valve implantation: alternative access options. Minerva Cardioangiol. 2013 Aug;61(4):429-35. PMID 23846009